CLINICAL TRIAL: NCT01827800
Title: New Media Obesity Treatment in Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0033
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: weight loss; primary care; eHealth
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eHealth weight loss intervention (Experimental): The 12-month eHealth behavioral intervention includes interactive self-monitoring and feedback, tailored skills training materials, telephone counseling calls from a study coach, and primary care provider counseling.
  Interventions: Behavioral: eHealth weight loss intervention
- Usual care (No Intervention): Participants in the usual care arm will receive the usual primary care services offered by their community health center primary care providers.

INTERVENTIONS:
Behavioral: eHealth weight loss intervention — This trial involves a multi-level, systems-change weight loss intervention. At the provider level, we make it easier for PCPs to deliver weight loss counseling by embedding patient progress data and counseling recommendations in the electronic health record. At the patient level, we provide engaging self-monitoring interfaces, immediate tailored feedback, skills training, and evidence-based lifestyle counseling from trusted care providers.
  Arms: eHealth weight loss intervention

SUMMARY:
This purpose of this trial is to determine whether a 12-month eHealth behavioral intervention that includes interactive self-monitoring and feedback, tailored skills training materials, telephone counseling calls, and primary care physician (PCP) counseling will produce greater weight change at 12 months than a standard primary care control.

DETAILED DESCRIPTION:
This is a patient randomized trial in which patients will be randomized into one of two treatment arms: 1) standard primary care; or 2) primary care plus a 12-month eHealth behavioral intervention (iOTA), which includes interactive self-monitoring and feedback, tailored skills training materials, 18 telephone counseling calls, and primary care provider counseling. The primary outcome is weight change at 12 months. Participants will be 351 adult male and female patients from local community health centers with obesity and a related comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 visit in the previous 12 months to an adult medicine, internal medicine, or family practice provider at a participating community health center
* BMI between 30.0-45.0 kg/m2 and weight ≤ 320 pounds
* Diagnosis of hypertension or diabetes

Exclusion Criteria:

* Current pregnancy
* Pregnancy in previous 12 months
* Heart attack/stroke in previous 2 years
* Active cancer diagnosis
* Current participation in another weight loss study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Weight change | Baseline - 12 months
  Weight will be measured at baseline and 12 months using a SECA 876 scale.

SECONDARY OUTCOMES:
The achievement and maintenance of > 5% weight loss | Baseline - 12 months
  Weight will be measured at baseline and 12 months using a SECA 876 scale.
Diet | Baseline - 12 months
  Dietary assessments will be performed at baseline and 12 months using the ASA24, a self-administered dietary recall measure developed by the National Cancer Institute.
Cardiometabolic risk markers | Baseline - 12 months
  Risk markers include waist circumference, systolic and diastolic blood pressure, lipid panel and A1c levels
Global Framingham risk score | Baseline - 12 months
  The Framingham Risk Score is a validated scoring system used to determine an individual's chances of developing cardiovascular disease. We will calculate this score at baseline and 12 months.
An evaluation of the intervention's impact and dissemination potential using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework | 12 and 24 months
  RE-AIM was originally developed as a framework for consistent reporting of research results and later used to organize reviews of the existing literature on health promotion and disease management in different settings. The acronym stands for Reach, Effectiveness, Adoption, Implementation, and Maintenance which together determine public health impact. More recently, RE-AIM has been used to translate research into practice and to help plan programs and improve their chances of working in "real-world" settings. The framework has also been used to understand the relative strengths and weaknesses of different approaches to health promotion and chronic disease self-management-such as in-person counseling, group education classes, telephone counseling, and internet resources.
Physical activity | Baseline -12 months
  Physical activity will be measured at baseline and 12 months using the GPAQ (the Global Physical Activity Questionnaire developed by the World Health Organization).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Gallis JA, Kusibab K, Egger JR, Olsen MK, Askew S, Steinberg DM, Bennett G. Can Electronic Health Records Validly Estimate the Effects of Health System Interventions Aimed at Controlling Body Weight? Obesity (Silver Spring). 2020 Nov;28(11):2107-2115. doi: 10.1002/oby.22958. Epub 2020 Sep 27. PMID 32985131
- [Derived] Steinberg D, Kay M, Burroughs J, Svetkey LP, Bennett GG. The Effect of a Digital Behavioral Weight Loss Intervention on Adherence to the Dietary Approaches to Stop Hypertension (DASH) Dietary Pattern in Medically Vulnerable Primary Care Patients: Results from a Randomized Controlled Trial. J Acad Nutr Diet. 2019 Apr;119(4):574-584. doi: 10.1016/j.jand.2018.12.011. PMID 30905430
- [Derived] McVay M, Steinberg D, Askew S, Bennett GG. Provider Counseling and Weight Loss Outcomes in a Primary Care-Based Digital Obesity Treatment. J Gen Intern Med. 2019 Jun;34(6):992-998. doi: 10.1007/s11606-019-04944-5. Epub 2019 Mar 19. PMID 30891688
- [Derived] Bennett GG, Steinberg D, Askew S, Levine E, Foley P, Batch BC, Svetkey LP, Bosworth HB, Puleo EM, Brewer A, DeVries A, Miranda H. Effectiveness of an App and Provider Counseling for Obesity Treatment in Primary Care. Am J Prev Med. 2018 Dec;55(6):777-786. doi: 10.1016/j.amepre.2018.07.005. Epub 2018 Oct 22. PMID 30361140
- [Derived] Foley P, Steinberg D, Levine E, Askew S, Batch BC, Puleo EM, Svetkey LP, Bosworth HB, DeVries A, Miranda H, Bennett GG. Track: A randomized controlled trial of a digital health obesity treatment intervention for medically vulnerable primary care patients. Contemp Clin Trials. 2016 May;48:12-20. doi: 10.1016/j.cct.2016.03.006. Epub 2016 Mar 17. PMID 26995281